## Effects of the ingestion of human, cow and modified cow milk, on glucose, amino acid and hormone responses in humans Acronym: PROLAT

## Statistical analysis

The statistical analysis was performed either on data absolute values, or as relative changes vs baseline. The incremental area(s) under the curve (iAUC) within specific time intervals were calculated using the trapezoidal approach. The one Way ANOVA was applied to analyze one single set of data in the four experimental groups, followed by post-hoc analysis using the Fisher's test. With multiple measurements over time, the data were analyzed using the two-Way Analysis of Variance (ANOVA) for repeated measurements, followed by the post-hoc Fisher's test. The two tailed Student's t test for unpaired data was used in some instances for head-to-head comparisons, as specifically indicated. The Statistica® Software (version 10) program was employed. A p value equal or less than 0.05 was considered statistically significant. Power analysis, sufficient to detect a  $\approx 30\%$  difference between two means, with a RMSSE (Root Mean Standardized Square Error) of <0.5, a power of 80%, and a two-sided level of significance of 0.05%, indicated a sample size of at least 29 subjects.